CLINICAL TRIAL: NCT00071734
Title: Brain Activation During Simple Vocal Behaviors
Status: Completed | Type: Observational
Sponsor: National Institute of Neurological Disorders and Stroke (NINDS) (NIH)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 040020; 04-N-0020
Record Dates: First submitted 2003-10-29; First posted 2003-10-29 (Estimated); Last update posted 2008-03-04 (Estimated); Status verified 2004-10

CONDITIONS: Auditory Perception
Keywords: fMRI; Auditory Feedback; Motor Control; Adult; BOLD; Healthy Volunteer; HV

SUMMARY:
This study will examine the central regions and brain activation patterns associated with simple vocal behaviors under conditions of normal auditory feedback-when people hear themselves speak. Such feedback plays a major role in learning and maintaining human voice control. But voice control can be harmed by neurological injury or disease, reducing the ability of a person to orally communicate. Research has shown that auditory feedback is continuously monitored, brought about by both automatic and voluntary corrections in the amplitude (loudness) and frequency of (pitch) of the human voice. This study aims to determine which areas of the brain have activity dependent on the level of blood oxygen. It will provide new knowledge about basic vocal motor control and provide a basis for investigations into the integration of hearing and speaking in human vocal expression throughout life.

Participants 18 to 45 years of age with normal hearing and voice function and with a steady heart rate may be eligible for this study.

Participants will be evaluated by a speech-language specialist, regarding a history of voice health and measures of voice function. They will be tested on their ability to vary voice amplitude and frequency and tested on their hearing. Also, they will undergo an electrocardiogram to determine their heart rate.

For the study, participants will undergo an MRI scan. During the MRI scan, patients will lie still on a table that can slide in and out of a metal cylinder surrounded by a strong magnetic field. Scanning time varies from 20 minutes to 3 hours, with most scans between 45 and 90 minutes. Patients may be asked to lie still for up to 90 minutes at a time. As the scanner takes pictures, there will be loud knocking noises, and patients will wear headphones to muffle the sound. The headphones will also enable patients to hear their voice. The patient's head will be positioned with a coil of 25 to 30 cm diameter and supported by a headrest. A microphone will be placed about 2 cm from the patient's mouth for communication and collection of data. Also, an angled mirror will be attached to the head coil, so that the patient can look outside of the scanner. By way of a projection screen, the patient will receive a visual cue to vocalize, or use his or her voice.

Patients will be asked to repeatedly do some of the following vocalization tasks: (1) rest, (2) hum or sigh without voicing (exhale), (3) hum or sigh audibly, (4) hum audibly while increasing or decreasing voice frequency, and (5) hum audibly while increasing or decreasing voice amplitude. During the scan, patients will be able to communicate with the MRI staff at all times and may ask to be moved out of the machine at any time. Some scans may be done in a 3 Tesla scanner. It is the latest advance in MRI, with a stronger magnetic field than in the more common 1.5 Tesla scanner. Functional MRI is done while a person is performing tasks, such as moving a limb or speaking. The fMRI scan will take about 1 hour.

DETAILED DESCRIPTION:
Auditory feedback plays a uniquely prominent role in the learning and maintenance of human voice control. Yet much of what is known about central voice motor control has come from research in non-human primates during production of genetically-determined vocalizations that do not rely upon auditory feedback. Extrapolation from studies of bat echolocation suggest that midbrain networks underlie automatic audiovocal error correction in humans; however, bats and humans differ greatly in anatomical and physiology.

ELIGIBILITY:
INCLUSION CRITERIA:

Males and females of any race or ethnicity will be eligible to participate in this study.

Volunteers must be between the ages of 18 and 45 with normal hearing and voice function. Participants will be further selected for having a steady heart rate. A history of voice training is not required, but participants must be able to produce grossly independent voice F0 and amplitude changes.

EXCLUSION CRITERIA:

Contraindications to participation include: pregnancy, cardiac pacemaker or auto defibrillator, artificial heart valve, neural pacemaker, surgical metal clips in the brain, eye, or on blood vessels, cochlear implants, ocular implants or foreign bodies such as metal shavings or splinters, insulin pump, implanted drug infusion device, shrapnel, bullet or shot wound, and tattooed makeup. Participants will be screened with the NMR Center Safety Screening Questionnaire which also includes items such as intraventricular shunts, transdermal medication patches, wire sutures, bone/joint pins, screws, nails, or plates, and body piercings. Given that surgical staples, orthopedic pins, orthodontic braces and dental implants are no longer considered absolute contraindications in MRI, Dr. Saxon or Dr. Kearney will approve or disapprove participation in the study based on their judgment of the MR compatibility of these items, using published guides including those referenced above.

Volunteers will be also excluded if they are found to be pregnant, report any tendency toward claustrophobia or are unable for any reason to lie still within an MR scanner.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 37
Dates: Start 2003-10; Study Completion 2004-10

CONTACTS AND LOCATIONS:
Locations (1):
- National Institute of Neurological Disorders and Stroke (NINDS), Bethesda, Maryland, United States

REFERENCES:
- [Background] Simonyan K, Jurgens U. Cortico-cortical projections of the motorcortical larynx area in the rhesus monkey. Brain Res. 2002 Sep 13;949(1-2):23-31. doi: 10.1016/s0006-8993(02)02960-8. PMID 12213296
- [Background] Gunji A, Hoshiyama M, Kakigi R. Identification of auditory evoked potentials of one's own voice. Clin Neurophysiol. 2000 Feb;111(2):214-9. doi: 10.1016/s1388-2457(99)00235-7. PMID 10680556
- [Background] Curio G, Neuloh G, Numminen J, Jousmaki V, Hari R. Speaking modifies voice-evoked activity in the human auditory cortex. Hum Brain Mapp. 2000 Apr;9(4):183-91. doi: 10.1002/(sici)1097-0193(200004)9:43.0.co;2-z. PMID 10770228